CLINICAL TRIAL: NCT00133432
Title: The Effect of Zinc Supplementation on Duration of Hospitalization in Tanzanian Children Presenting With Acute Pneumonia
Brief Title: Zinc and Pneumonia Protocol
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 03-179; NCT00197717 (obsolete NCT alias)
Record Dates: First submitted 2005-08-19; First posted 2005-08-23 (Estimated); Last update posted 2019-01-29 (Actual); Status verified 2010-03

CONDITIONS: Respiratory Infections, Acute
Keywords: Pneumonia, acute respiratory infections, zinc, Tanzania, children, infants, hospitalization
MeSH Terms: conditions — Respiratory Tract Infections; Pneumonia | interventions — Zinc

INTERVENTIONS:
Drug: Zinc

SUMMARY:
Undernutrition in children less than five years of age is common throughout sub-Saharan Africa. Nutritional deficiencies may lead to less ability to fight infectious diseases. The purpose of this study is to determine whether zinc supplements plus standard antibiotics reduce the length of hospitalization in children with pneumonia. Six hundred children aged 6-36 months diagnosed with pneumonia and admitted to Muhimbili National Hospital (MNH), Dar es Salaam, Tanzania, will participate in this study. Half of the children will receive daily supplements of zinc, and the other half will receive placebo tablets (dummy pills containing no medication). Each child will be followed for 6 weeks after hospital discharge to check for recovery from the illness. All children in both groups will receive antibiotics and supportive care to manage pneumonia, according to the standards of care at MNH and Amana Municipal Hospital in accordance with the Recommendations of the Ministry of Health, Tanzania.

DETAILED DESCRIPTION:
Undernutrition in children less than five years of age is prevalent throughout sub-Saharan Africa and is often associated with multiple micronutrient deficiencies, such as vitamin A and zinc. These deficiencies are probably a reflection of the poverty and poor living conditions that contribute to the lack of proper nutrition. The potential adverse effect of even subclinical deficiency in various micronutrients (including zinc) on optimal physiological function may lead to an exacerbation of infectious diseases in children living in these parts of the world. The primary objective of this randomized, double-blind, placebo-controlled study is to determine whether oral zinc supplementation plus standard antibiotics significantly alters the duration of required hospitalization in children with radiologically confirmed acute pneumonia. Six hundred children aged six months to 36 months diagnosed with radiologically confirmed acute pneumonia and admitted in the general pediatric wards of Muhimbili National Hospital (MNH), Dar es Salaam, Tanzania, will be recruited. Upon enrollment, half of the subjects will receive daily oral supplements of 25 mg of elemental zinc and the control group will receive placebo tablets. Children randomized to receive zinc supplements will be given a daily dose of 25 mL of reconstituted solution from effervescent tablets equivalent to 25 mg of elemental zinc in two divided doses (12.5 mg twice daily) by a study coordinator during the hospital phase of treatment for pneumonia. Children randomized to the control group will receive placebo effervescent tablets identical in taste and appearance to those tablets containing zinc. Compliance to the regimen will be directly observed by the study coordinator, and clinical response will be closely monitored throughout hospital stay. Each child will be followed for six weeks after hospital discharge to assess for recovery from the illness. All children in both groups will receive antibiotics and supportive care to manage pneumonia, as deemed appropriate according to the standards of care as practiced at MNH and Amana Municipal Hospital in accordance with the Recommendations of the Ministry of Health, Tanzania.

ELIGIBILITY:
Inclusion Criteria:

1. Age six months to 36 months inclusive.
2. A primary clinical diagnosis of acute pneumonia, which consists of a child presenting with cough or difficulty breathing with the following features:

   1. Tachypnea: Respiratory rate greater than or equal to 50 breaths per minute for children aged 6 months up to 12 months and greater than or equal to 40 breaths per minute for children aged 12 months to 36 months.
   2. Fever: Temperature greater than or equal to 37.5 degrees Celsius with an axillary thermometer.
   3. Any one of the following signs: Flaring of alae nasi, visible indrawing of the lower chest wall muscles on inspiration, central cyanosis, inability to feed, lethargy, or crepitations, i.e. short crackling noises heard during the inspiratory phase of respiration.
3. Chest x-ray abnormalities consistent with an inflammatory process such as distinctly confined dense abnormality or large pleural effusion (i.e. pneumonia or lower respiratory tract infection), not just any change such as pulmonary edema.
4. Parent/caregiver willing to give informed consent and to allow HIV testing of their child.
5. Child able to take study regimen (zinc supplement/placebo).
6. Parents/caregivers willing to comply with a follow-up study visit.
7. Child is anticipated to survive the episode of pneumonia and has no other serious concomitant medical condition that would affect their ability to survive the acute episode of pneumonia.

Exclusion Criteria:

1. Presence of severe malnutrition according to Wellcome Classification (marasmus, marasmic-kwashiorkor, and kwashiorkor), which requires microniutrient supplementation including zinc or any other sign of severe malnutrition.
2. Prior known or current diagnosis of full blown AIDS meeting World Health Organization clinical case definition. Children who are only HIV-positive and have acute pneumonia will not be excluded from the study.
3. Subjects with active tuberculosis.
4. Subjects with active measles.
5. Subjects with known or suspected signs of systemic illness (e.g. sepsis, acute meningitis, hemodynamic instability).
6. Subjects with diarrhea defined as passage of 3 or more loose or watery stools in the past 24 hours.
7. Subjects for which the number of days of illness prior to admission is greater than 3 days.
8. Known intolerance or allergy to zinc or zinc-containing products.
9. Subjects presently receiving zinc supplementation.

Ages: 6 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 600
Dates: Start 2005-09

CONTACTS AND LOCATIONS:
Locations (1):
- Muhimbili University, College of Health Sciences, Dar es Salaam, Tanzania